CLINICAL TRIAL: NCT04112602
Title: Respiratory Impairment in Mucopolysaccharidosis Patients: Impact of Glycosaminoglycans (GAG) on the Proteases/Antiproteases Balance
Brief Title: Respiratory Cathepsins, Proteases Inhibitors and Glycosaminoglycans (GAG) in Mucopolysaccharidosis
Acronym: RespiGAG
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI19/RespiGAG; 2019-A01361-56 (Other: IdRCB); 19.05.17.43323 RIPH 3 HPS (Other: CPP)
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Mucopolysaccharidoses
Keywords: mucopolysaccharidosis; lung cathepsins; proteases inhibitors; glycosaminoglycans
MeSH Terms: conditions — Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pulmonary samples (sputum / tracheal aspiration)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with MPS: In this cohort are included patients under 18 years old with MPS (all types). The objective is to be representative of the diversity of MPS, and of this evolution.
  Interventions: Other: Sputum; Other: Tracheal aspiration
- Non-MPS patients: In this control group are included patients under 18 years old, with no respiratory problems, no MPS.
  Interventions: Other: Tracheal aspiration

INTERVENTIONS:
Other: Sputum — Sputum will be collected after a respiratory physiotherapy session, scheduled as part of routine care.
  Groups: Patients with MPS
Other: Tracheal aspiration — Tracheal aspirations will be collected in intubated patients (intubation for surgery under general anesthesia).

SUMMARY:
Mucopolysaccharidosis (MPS) are a group of inherited, metabolic diseases caused by a deficiency of lysosomal enzymes that degrade glycosaminoglycans (GAGs). Loss of their activity results in cellular accumulation of GAGs fragments leading to progressive multi-system manifestations, with respiratory impairment. The cellular and molecular mechanisms responsible for the pulmonary impairment remain largely unknown. Specific GAGs, such as those accumulating in MPS, may act as potent inhibitors of some respiratory enzymes, like lysosomal cathepsins, depending on the nature of GAGs and their concentration. It is well established that deregulation of cathepsins levels plays a major role in the pathophysiology of some chronic respiratory diseases, such as cystic fibrosis. The role of cathepsins and their inhibitors in respiratory samples of MPS patients has never been studied. This study will focus on the status/activity of these proteases and their endogenous inhibitors in the sputum or tracheal aspiration of patients with MPS. Our main hypothesis is that high levels of GAGs in MPS patients impair the physiological activity of cathepsins and their inhibitors.

DETAILED DESCRIPTION:
Mucopolysaccharidosis (MPS) are a group of inherited, metabolic diseases caused by a deficiency of lysosomal enzymes that degrade glycosaminoglycans (GAGs). Loss of their activity results in cellular accumulation of GAGs fragments leading to progressive multi-system manifestations (central nervous system involvement, dysmorphism, skeletal abnormalities, cardiomyopathy, ear/nose/throat and respiratory problems). Impairment of pulmonary function is an important health problem for patients with MPS.

Various therapeutic approaches have been developed to restore deficient enzymatic activity (stem cell transplantation, enzyme replacement therapy, gene therapy), but new therapeutic approaches may be required, in addition to these current conventional treatments. In particular, respiratory failure is not fully restored. The cellular and molecular mechanisms responsible for lung dysfunction remain today largely unknown and require additional investigations. It is well established that GAGs, upon specific conditions either stimulate or inhibit the activity of specific enzymes named cathepsins.

Cysteine cathepsins are lysosomal proteases that can be secreted extracellularly by macrophages, epithelial cells and fibroblasts. Imbalance between cathepsins and their inhibitors in favor to proteolysis has been demonstrated in patients with chronic pulmonary diseases (silicosis, cystic fibrosis). By contrast, high levels of their endogenous inhibitors are found in idiopathic fibrosis. Interestingly, previous studies reported that accumulation of sulphated GAGs (chondroitin sulfate, heparan sulfate, dermatan sulfate) impaired the collagenolytic activity of cathepsin K in a MPS I mouse model, supporting that cathepsin K participates to the pathophysiology of the bone involvement in patients with MPS. Moreover, other related cathepsins are regulated in vitro by GAGs.

Thus, inhibition of cathepsins may contribute to the respiratory impairment in MPS patients. However, their expression and their role in the airway of MPS patients are still unknown. Moreover, little is known on GAG levels in MPS lungs. The main hypothesis of the proposed research is to evaluate the levels of sulfated GAGs (heparan sulfate, chondroitin sulfate, dermatan sulfate) in respiratory samples of MPS patients and the ability of theses GAGs to modulate the proteolytic activities of lysosomal cathepsins. This would lead to an abnormal remodeling of the extracellular matrix architecture, contributing to the respiratory disorders of patients with MPS. To validate this hypothesis, a correlational study will be performed to find a relationship between cathepsins expression/activity, GAGs concentrations and respiratory function.

This is a multicentre, prospective, non-interventional and case-control study (patients with MPS vs non-MPS patients). Pulmonary samples (biological waste) will be collected in patients after either a respiratory physiotherapy session (scheduled for routine care) or by tracheal aspiration when patients are intubated (intubation for imaging or surgery under general anesthesia). Collected samples will be used to assess the level of expression and activity of cathepsins and their inhibitors and the amount of sulfated GAGs.

Patients with MPS will be recruited in some Reference and Competence Centers for Metabolic Diseases in France (Angers, Bordeaux, Brest, Rennes, Toulouse, Tours). The non-MPS patients will be recruited at the Tours University Hospital (Pediatric Resuscitation).

Some medical data of patients with MPS will be collected retrospectively from the medical record. These data will be age, sex, type of MPS, respiratory assessment.

The data collected for the non-MPS patients will be age and sex.

The expected benefits are:

1. Better understanding of the respiratory pathophysiology in MPS patients: by understanding the molecular cathepsins/GAGs interactions.
2. Development of new therapeutic approaches for respiratory disease in patients with MPS:

   If we can prove that there is a dysregulation of pulmonary cathepsin activity in patients with MPS, a treatment that will restore this activity would be of great interest. This type of treatment is already studied in bone diseases such as osteoporosis. This treatment would be complementary to current conventional therapies, like stem cell transplant or enzyme replacement therapy.
3. New therapeutic approaches potentially effective for other problems in patients with MPS:

The mechanism of cathepsin activity inhibition by GAGs is probably not lung-specific. GAGs accumulation and cathepsin expression are ubiquitous in humans. The role of cathepsins dysregulation by GAGs has already been described to explain some bone or cardiac involvements. These new therapeutic approaches could therefore also have a beneficial effect on other organs involvement in patients with MPS.

ELIGIBILITY:
Patients with MPS:

Inclusion Criteria:

* Patient with a confirmed diagnosis (enzymatic activity, and/or genotyping) of MPS, all types (I, II, III, IV, VI, VII, IX)
* Aged from 0 to 17 years old

Non inclusion Criteria:

* Chronic respiratory disease independent of MPS disease (potential interferences with our analyzes)
* Inability to obtain pulmonary samples
* Refusal of the patient, parent or legal representative to participate in this study

Exclusion Criteria:

* Impossibility to use pulmonary samples (insufficient volume, conservation problem, etc.)

Non-MPS patients:

Inclusion Criteria:

* Patient with no respiratory disease
* Aged from 0 to 17 years old

Non inclusion Criteria:

* Emergency medical situation
* Inability to obtain pulmonary expectoration
* Refusal of the patient, parent or legal representative to participate in this study

Exclusion Criteria:

* Impossibility to use pulmonary samples (insufficient volume, conservation problem, etc.)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with MPS:
  In this cohort are included patients under 18 years old with MPS (all types). The objective is to be representative of the diversity of MPS, and of this evolution.
  Non-MPS patients:
  In this control group are included patients under 18 years old, with no respiratory problems, no MPS.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of the expression of pulmonary cathepsins, proteases inhibitors and GAGs in MPS patients. | Day 1
  Detection and identification by Western blot. Results will be compared to non-MPS patients.
Quantification of pulmonary cathepsins, protease inhibitors and GAGs in MPS patients. | Day 1
  Quantification by kinetics and ELISA assays. Results will be compared to non-MPS patients.

SECONDARY OUTCOMES:
Pulmonary cathepsins enzymatic activity measurement. | Day 1
  Enzyme activity measurement by enzymatic kinetics techniques.

CONTACTS AND LOCATIONS:
Overall Officials: François Labarthe, MD-PhD, Study Director — University Hospital, Tours
Locations (7):
- France (7):
  - Metabolic Disease Competence Centre - Medical Genetics Department - University Hospital, Angers, Angers
  - Metabolic Disease Reference Centre - Medical Genetics Department - University Hospital, Bordeaux, Bordeaux
  - Metabolic Disease Competence Centre - Medical Genetics Department - University Hospital, Brest, Brest
  - Metabolic Disease Competence Centre - Pediatrics Department - University Hospital, Rennes, Rennes
  - Metabolic Disease Reference Centre - Pediatrics Department - University Hospital, Toulouse, Toulouse
  - Metabolic Disease Reference Centre - Pediatrics Department - University Hospital, Tours, Tours
  - Pediatric Resuscitation Unit - Universty Hospital, Tours, Tours

REFERENCES:
- [Background] Khan SA, Peracha H, Ballhausen D, Wiesbauer A, Rohrbach M, Gautschi M, Mason RW, Giugliani R, Suzuki Y, Orii KE, Orii T, Tomatsu S. Epidemiology of mucopolysaccharidoses. Mol Genet Metab. 2017 Jul;121(3):227-240. doi: 10.1016/j.ymgme.2017.05.016. Epub 2017 May 26. PMID 28595941
- [Background] Rapoport DM, Mitchell JJ. Pathophysiology, evaluation, and management of sleep disorders in the mucopolysaccharidoses. Mol Genet Metab. 2017 Dec;122S:49-54. doi: 10.1016/j.ymgme.2017.08.008. Epub 2017 Aug 25. PMID 28964643
- [Background] Kobayashi H. Recent trends in mucopolysaccharidosis research. J Hum Genet. 2019 Feb;64(2):127-137. doi: 10.1038/s10038-018-0534-8. Epub 2018 Nov 19. PMID 30451936
- [Background] Wilson S, Hashamiyan S, Clarke L, Saftig P, Mort J, Dejica VM, Bromme D. Glycosaminoglycan-mediated loss of cathepsin K collagenolytic activity in MPS I contributes to osteoclast and growth plate abnormalities. Am J Pathol. 2009 Nov;175(5):2053-62. doi: 10.2353/ajpath.2009.090211. Epub 2009 Oct 15. PMID 19834056
- [Background] Lalmanach G, Saidi A, Marchand-Adam S, Lecaille F, Kasabova M. Cysteine cathepsins and cystatins: from ancillary tasks to prominent status in lung diseases. Biol Chem. 2015 Feb;396(2):111-30. doi: 10.1515/hsz-2014-0210. PMID 25178906
- [Background] Bromme D, Lecaille F. Cathepsin K inhibitors for osteoporosis and potential off-target effects. Expert Opin Investig Drugs. 2009 May;18(5):585-600. doi: 10.1517/13543780902832661. PMID 19388876
- [Background] Baldo G, Tavares AM, Gonzalez E, Poletto E, Mayer FQ, Matte UD, Giugliani R. Progressive heart disease in mucopolysaccharidosis type I mice may be mediated by increased cathepsin B activity. Cardiovasc Pathol. 2017 Mar-Apr;27:45-50. doi: 10.1016/j.carpath.2017.01.001. Epub 2017 Jan 6. PMID 28104572
- [Background] Sage J, Mallevre F, Barbarin-Costes F, Samsonov SA, Gehrcke JP, Pisabarro MT, Perrier E, Schnebert S, Roget A, Livache T, Nizard C, Lalmanach G, Lecaille F. Binding of chondroitin 4-sulfate to cathepsin S regulates its enzymatic activity. Biochemistry. 2013 Sep 17;52(37):6487-98. doi: 10.1021/bi400925g. Epub 2013 Sep 4. PMID 23968158
- [Background] Kubaski F, Tomatsu S, Patel P, Shimada T, Xie L, Yasuda E, Mason R, Mackenzie WG, Theroux M, Bober MB, Oldham HM, Orii T, Shaffer TH. Non-invasive pulmonary function test on Morquio patients. Mol Genet Metab. 2015 Aug;115(4):186-92. doi: 10.1016/j.ymgme.2015.06.007. Epub 2015 Jun 23. PMID 26116954